CLINICAL TRIAL: NCT00294281
Title: A Pilot Study to Assess the Tolerability and Exploratory Efficacy of Vagus Nerve Stimulation (VNS) Using the VNS Therapy System in Patients With Refractory Fibromyalgia With and Without Major Depression
Brief Title: Vagus Nerve Stimulation for Treating Adults With Severe Fibromyalgia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Gudrun Lange, PhD, University of Medicine and Dentistry of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01AR053732 (NIH); 5R01AR053732 (NIH); FM-01
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2010-07

CONDITIONS: Fibromyalgia
Keywords: Pain; Tenderness; Depression; Work Disability; Physical Function; Quality of Life; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Pain; Depression; Chronic Pain | interventions — Vagus Nerve Stimulation; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Participants will undergo surgical implantation of the VNS system. This will be followed by a 2-week recovery period, then a 2-week period of gradually increasing the electrical output of the VNS system, and finally a 12-week VNS treatment period during which the electrical output level will remain constant. Follow-up will occur until Month 24.
  Interventions: Device: Vagus Nerve Stimulation (VNS) Therapy

INTERVENTIONS:
Device: Vagus Nerve Stimulation (VNS) Therapy — The VNS Therapy System Pulse Generator is an implantable, multi-programmable bipolar pulse generator. The pulse generator will deliver electrical signals to the vagus nerve via bipolar leads. A programming wand and software system enable non-invasive programming, functional assessments, interrogation, and data retrieval.

SUMMARY:
Fibromyalgia syndrome (FMS) is a long-term disorder that is characterized by widespread body pain and tender points in joints, muscles, tendons, and other soft tissues. Other symptoms associated with the disorder include fatigue and depression. The cause of FMS is unknown, and conventional treatments are often unsuccessful in adequately relieving pain. For people with severe, unrelenting pain, which is referred to as refractory FMS, opioid maintenance therapy may be an option, but it comes with the dangerous potential of addiction and is therefore avoided if possible. Vagus nerve stimulation (VNS), in which a nerve located in the neck receives electrical input, may be an option for providing pain relief. The purpose of this study is to determine the safety, tolerability, and effectiveness of VNS as a treatment for people with refractory FMS.

DETAILED DESCRIPTION:
FMS affects about 5% of the general population and occurs most often in women between the ages of 20 and 50 years old. Overall, more than 80% of FMS patients report that pain is the primary symptom that limits their ability to work, about 30% of patients are disabled, and about 45% collect Social Security Disability insurance. Conventional treatments, which include pharmacological and behavioral interventions, fail to provide adequate pain relief in more than half of FMS patients, strongly suggesting the need for improved treatment options.

One such option is a treatment called vagus nerve stimulation (VNS), in which short bursts of electrical energy are directed into the brain by way of the vagus nerve. The vagus nerve is a cranial nerve that originates in the brainstem, travels through the neck, and then continues down through the thorax and abdomen. The nerve acts as both a sensory and motor nerve, and it can regulate several brain areas involved in pain and emotional processing. With VNS, a small battery device is surgically implanted under the skin, usually under the chest, and provides the necessary electrical energy for stimulation. Although VNS has been FDA approved for some forms of epilepsy and depression, it has yet to receive FDA approval for FMS. Also, it is unknown whether the safety and tolerability profile of an FMS patient receiving VNS is the same as that of a patient with epilepsy or depression who is receiving VNS. The purpose of this study is to determine the safety, tolerability, and effectiveness of VNS as a treatment option for adults with refractory FMS.

Participants will be in this study for about 25 months. An initial screening period that may last up to 6 weeks will include a medical history review, various examinations, and the use of a wrist-mounted device called an Actiwatch to record pain severity and mood over seven consecutive days. Eligible participants will then undergo surgical implantation of the VNS system. This will be followed by a 2-week recovery period, then a 2-week period of gradually increasing the electrical output of the VNS system, and finally a 12-week VNS treatment period during which the electrical output level will remain constant, unless a participant develops intolerable side effects. Study visits will occur weekly for the first month after implantation and then every 2 weeks during the treatment period. During most study visits, participants will undergo a clinical assessment, including evaluation of any side effects, and they will complete written assessments on pain, mood, fatigue, and quality of life and sleep. The VNS system will also be checked for safety and programmed appropriately. During the Week 16 visit, some of the screening evaluations will be repeated. Also at Week 16, which will mark the end of the treatment period, participants will have the option to continue receiving treatment. All participants will have follow-up evaluations at Months 6, 9, 12, and 24. Participants who wish to retain the VNS implantation beyond the length of the study will be referred to a qualified neurologist for follow-up care. For the other participants, the VNS system will be turned off and surgically explanted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FMS for at least 2 years, as according to the 1990 guidelines of the American College of Rheumatology (ACR) criteria. In addition, ruling out of any other medical illness to which pain may be attributed.
* Inadequate relief in FMS pain despite good treatment efforts using standard pharmacological pain management. Only patients who are work-disabled because of FMS pain are eligible for study participation if they are on opioid maintenance therapy.
* Overall FMS pain at an intensity of 5 or greater on a 0-10 verbally anchored pain intensity scale, on more than 50% of days over a consecutive 7-day period before study entry
* Has not changed pharmacological and/or non-pharmacological (e.g., yoga, exercise) treatment regimen for the 4 weeks before the first study visit and continues to experience severe pain
* At least average premorbid IQ, as assessed by the vocabulary subtest of the WAIS-III, which is a standardized, well-validated index of premorbid intellectual function
* Willing to use an acceptable method of birth control
* Able to comply with all testing and follow-up visit requirements defined by the study protocol
* Currently lives within a 2-hour driving commute to the study site

Exclusion Criteria:

* Rheumatologic condition other than FMS
* Secondary FMS, in which FMS is comorbid with another rheumatologic condition
* Reports that FMS pain began after a physical trauma
* In litigation that is associated with FMS condition at study entry
* Severe lifetime or current diagnosis of psychotic depression, bipolar disorder, schizophrenia, schizoaffective disorder, or other psychotic disorders or has a clear history of other psychiatric illness before the onset of FMS
* Diagnosed with major depressive disorder and has attempted to commit suicide in the past or has active suicidal ideation
* Lifetime or current history of dependence or abuse of pain medication or alcohol
* Treatment with an antipsychotic drug within 3 months of study entry
* Demonstrated a known placebo response in a previous study
* Treatment with botulinum toxin or local steroid injection for FMS within 2 months of study entry
* History of myocardial infarction or cardiac arrest
* Received general anesthesia within 30 days of implantation surgery
* Treatment with an investigational drug within a clearance duration of five times the half-life of the investigational drug or within 4 weeks of study entry
* Currently using another investigational device or drug
* Significant heart or lung condition currently under treatment and resulting in an American Society of Anesthesiologists (ASA) score greater than III
* Unilateral or bilateral cervical vagotomy
* Demand cardiac pacemaker, implantable defibrillator, or other implantable stimulator
* Any of the following conditions if over the age of 50 years old: cardiac conductance abnormalities, Wolf-Parkinson-White Syndrome, surgical intervention for bradycardia, history of prolonged QT interval, or a history of syncopal or pre-syncopal episodes
* Likely to require a whole body MRI after VNS system implantation
* Currently receiving or likely to receive after implantation short-wave diathermy, microwave diathermy, or therapeutic ultrasound diathermy
* Plans to relocate or move to a location distant from the study site within 1 year of study entry
* Previously enrolled in this or any other VNS system study
* Pregnant

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2006-10; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Measured at Week 16, which is the acute study exit

SECONDARY OUTCOMES:
FM 20 multidimensional response index (FM 20) | Measured at Week 16, which is the acute study exit
Assessment of pain intensity | Measured at Week 16, which is the acute study exit
Assessment of function | Measured at Week 16, which is the acute study exit
Assessment of patient global perception | Measured at Week 16, which is the acute study exit

CONTACTS AND LOCATIONS:
Overall Officials: Gudrun Lange, PhD, Principal Investigator — University of Medicine and Dentistry of New Jersey
Locations (1):
- University of Medicine and Dentistry of New Jersey, Newark, New Jersey, United States

REFERENCES:
- [Derived] Lange G, Janal MN, Maniker A, Fitzgibbons J, Fobler M, Cook D, Natelson BH. Safety and efficacy of vagus nerve stimulation in fibromyalgia: a phase I/II proof of concept trial. Pain Med. 2011 Sep;12(9):1406-13. doi: 10.1111/j.1526-4637.2011.01203.x. Epub 2011 Aug 3. PMID 21812908